CLINICAL TRIAL: NCT03683199
Title: Objective Assessment for Cleft Lip Nasal Deformity Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hafsa Gamal Muhammad bakheet, Assistant teacher, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUH
Record Dates: First submitted 2018-09-11; First posted 2018-09-25 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Nose; Anomaly
Keywords: Secondary; Cleft; Lip; Nose; Deformity; Correction; Objective; Assessment
MeSH Terms: conditions — Congenital Abnormalities; Neoplasm Metastasis; Lymphoid Interstitial Pneumonia | interventions — Rhinoplasty

STUDY DESIGN:
Intervention Model Description: The total sample size will be 27 patients to study as calculated using G power version 3.1.3, in order to detect a significant difference in the mean of nasal ratios before and after surgery in the studied group (one of basic tools to measure the outcome). Assumed Effect size= 0.5, Power =0.80, Alpha error = 0.05.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cleft lip nasal deformity (Experimental): •Anthropometric evaluation of the nose (will be measured pre and post-operative) This represents the objective evaluation. It will be done by measuring the angles and ratios of the nose and its relation to the face. Common parameters will be measured from the photos (frontal, oblique, lateral and basal views) for all the patients to compare the pre-operative measures with the post-operative ones.
  MSCT flesh mode will be used to measure nose related angels and ratios. It also gives idea about nasal skeleton pre-operative for proper design of the operative strategy, and it will be done post-operative for assessment and comparizon.
  Interventions: Procedure: Rhinoplasty

INTERVENTIONS:
Procedure: Rhinoplasty — The cleft lip rhinoplasty will be performed under general anesthesia.
  1: 100,000 epinephrine will be infiltrated in the columellar incision and in the septum.
  Open approach rhinoplasty will be used. A step ladder incision placed at the patient's columella, and continued with infra-cartilaginous incision.
  The columellar skin flap along with the nasal tip skin will be dissected from the lower lateral cartilages.
  Harvesting of the septal cartilage, to be used as spreader graft and columellar graft. Correction of the septal deviation.
  Lengthening of the columella on the expense of the ala. Correction of the nasal tip by suturing techniques and by cartilage grafts.

SUMMARY:
Rhinoplasty remains one of the most challenging procedures in plastic surgery, and patients with cleft lip nasal deformity pose an even greater challenge, in which biggest issue is to achieve caudal nose harmony and creation of symmetrical nostrils with patent normal nasal function

DETAILED DESCRIPTION:
Cleft lip and palate represent the most common birth defects affecting the head and neck region. It has been estimated, based on global birth rates that a child born with a cleft every 2.5 minutes .which is associated with varying degrees of nasal deformity grading from mild to severe inadequate function, shape and appearance of the nose. Functional impairment of the nose has been reported in 70% of cases with cleft lip. It negatively affects patients' personal and professional lives, physical activity, well-being and general quality of life.

However, historical interest in cleft lip and palate was traced to pre-Columbian artisan; the interest in the associated nasal deformities only began with rhinoplasty techniques introduced in the 19th century. That's why despite the great improvement achieved in primary repair of cleft lip and nasal deformity, the secondary cleft and nasal deformity still occur in significant number of patients, and the surgical management of the nasal deformity remains a functional and aesthetic dilemma for patients, their families and for reconstructive surgeons.

Lake of objective assessment of the initial severity and the changes introduced by growth and by surgical treatment lead to inability to optimize a treatment of cleft lip nasal deformity, hence there is no perfect surgical technique exists and surgeons must tailor approaches to individuals and evolve techniques to best serve each patient.

Although surgery can give dramatic effect, the lack of objective assessment of different surgical procedures results in decision that is based on the experience of the surgeon.

Secondary rhinoplasty is done after facial growth is completed. This is around 14 to 16 years old in female patients and 16 to 18 years old in male patients. Surgical techniques rely on well-accepted open rhinoplasty principles and are applied for unilateral or bilateral cleft nasal deformities.

Careful complete analysis followed by logical plan for each case is the key stone for success.

Multislice CT Flesh mode will be used for measuring some angles and ratios of the nose and its relation to the face. The results will be recorded at the spread sheet and the preoperative and post operative results will be compared. Other parameters can also be measured, as long as user records the measurements manually.

ELIGIBILITY:
Inclusion Criteria:

1. Age group: > 14-16 years old females and >16-18 years old male patients.
2. Patients with unilateral or bilateral cleft lip nasal deformity that isn't previously operated.

Exclusion Criteria:

1. Previous rhinoplasty operated CLND cases.
2. Patients who need skeletal base reconstruction.
3. Syndromic cases.
4. Post traumatic nasal deformity.
5. Female patients less than 14 years' old and male patients less than 16 years old.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — 1- Age group: > 14-16 years old females and >16-18 years old male patients
Enrollment: 1 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
Objective Assessment for cleft lip nasal deformity correction using MSCT with 3Dimentions in flesh mode (to compare some nasal lengths in millimeters before and after correction) | three years
  we will use Multislice CT 3D flesh mode to compare the columellar length in millimeters and inter-alar dimensions in millimeters before and after the surgical correction
Objective Assessment for cleft lip nasal deformity correction using MSCT with 3Dimentions in flesh mode (to compare some nasal lengths in millimeters before and after correction) | three years
  Using MSCT with 3Dimentions in flesh mode, we will compare the angle of sepal deviation in degrees, before and after cleft nose rhinoplasty

SECONDARY OUTCOMES:
Patient's subjective assessment pre and post-operative using Rhinoplasty Outcome Evaluation questionnaire | three years
  Patient will be asked to answer six simple questions to assess his physical, mental / emotional and social life. These questions are:
  How well do you like the appearance of your nose? How well are you able to breathe through your nose? How much do you feel your friend and loved ones like your nose? How much do you feel your friend and loved ones like your nose? Do you think your current nasal appearance limits your social and professional activities? How confident are you that your nasal appearance is the best can be? Patients will give answer to those questions as: not at all (0) somewhat (1) moderately (2) very much (3) completely (4) In order to reach the final result in the scale, we will add the responses from each question, and such result will be divided by 24 and multiplied by 100.
  The final result will then be divided in classes, according to quartiles: zero to <25 and 25 to <50 (failure); 50 to <75 (good); and ≥75 (excellent).

CONTACTS AND LOCATIONS:
Locations (1):
- Hafsa gamal, Asyut, Egypt